CLINICAL TRIAL: NCT01757262
Title: Safety and P2Y12 Receptor Inhibition Effects of Ticagrelor and Clopidogrel in Vietnamese Patients With Coronary Heart Disease: A Randomized, Open Label, Crossover Study
Brief Title: A Clinical Study of Safety and P2Y12 Receptor Inhibition Effects of Ticagrelor and Clopidogrel in Vietnamese Patient
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D5130C00078
Record Dates: First submitted 2012-12-21; First posted 2012-12-28 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Ticagrelor; Clopidogrel

ARMS (2):
- Ticagrelor (Experimental): 90 mg Ticagrelor
  Interventions: Drug: 90 mg Ticagrelor
- Clopidogrel (Active Comparator): 75mg Clopidogrel
  Interventions: Drug: 75mg Clopidogrel

INTERVENTIONS:
Drug: 90 mg Ticagrelor — Morning and Evening dose for 5 days
  Arms: Ticagrelor
Drug: 75mg Clopidogrel — Morning dose for 5 days
  Arms: Clopidogrel

SUMMARY:
Study in Vietnamese Patients with Coronary Heart Disease to investigate safety and P2Y12 Receptor Inhibition Effects of Ticagrelor and Clopidogrel

DETAILED DESCRIPTION:
Safety and P2Y12 Receptor Inhibition Effects of Ticagrelor and Clopidogrel in Vietnamese Patients with Coronary Heart Disease: A Randomized, Open Label, Crossover Study

ELIGIBILITY:
Inclusion Criteria:

* Male or female Vietnamese patients (as confirmed by the Principal Investigator) aged >18 years with suitable veins for cannulations or repeated venipunctures and stable coronary heart disease
* Stable use of aspirin 75 to 100 mg daily for at least the preceding 2 weeks and which will be continued throughout the study period
* Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive
* Women must have a negative urine pregnancy test at Visit 1

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study
* Unstable angina or any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IP
* Patients who had acute coronary syndrome or stent placed within 12 months of screening
* Planned arterial revascularization
* Current use of ADP receptor blockers (eg, clopidogrel, ticlopidine, prasugrel), dipyridamole or cilostazol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamics of Ticagrelor on P2Y12 receptor blockade measured by the VerifyNow P2Y12 assay[expressed as P2Y12 reaction units (PRU)] | Day 1 pre-dose and at 0 (pre-dose), 1, 2, 8, 12 and 24 hours post morning dose on Day 5
Pharmacodynamics of Clopidogrel P2Y12 receptor blockade measured by the VerifyNow P2Y12 assay[expressed as P2Y12 reaction units (PRU)] | Day 1 pre-dose and at 0 (pre-dose), 1, 2, 8, 12 and 24 hours post morning dose on Day 5

SECONDARY OUTCOMES:
Safety profile in terms of adverse events, blood pressure, pulse, ECG (Electrocardiogram), physical examination, and safety laboratory variables | From screening to followup (8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen Lan Viet, MD, Principal Investigator — National Heart Institute, Bach Mai Hospital, Vietnam; Judith Hsia, MD, Study Director — Astrazeneca, Wilmington, US; Miriana Kujacic, MD, Study Chair — Astrazeneca, Molndal, Sweden